CLINICAL TRIAL: NCT06753318
Title: Validation of a Multimodal Artificial Intelligence Model in in Diagnosing Pancreatic Solid Lesions: a Prospective, Multicenter, Randomized, Controlled Trial
Brief Title: Validation of Joint-AI in Diagnosing Pancreatic Solid Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Beijing Union Hosptial (Unknown); Affiliated Drum Tower Hospital of Nanjing University Medical School (Unknown); Shanghai Longhua Hospital (Unknown); Beijing Friendship Hospital (Other); Qilu Hospital of Shandong University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Bin Cheng, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Joint-AI 2024
Record Dates: First submitted 2024-12-17; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer; Pancreatitis; Pancreatic Neuroendocine Neoplasms (pNETs); Autoimmune Pancreatitis; Solid Pseudopapillary Neoplasm of the Pancreas
Keywords: pancreatic cancer; artificial intelligence; endoscopic ultrasound
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis; Autoimmune Pancreatitis

STUDY DESIGN:
Intervention Model Description: 1. First, participants are randomized into three parallel groups: conventional diagnosis group, Joint-AI assistance group, and Interpretable Joint-AI assistance group.
  2. For participants within the Joint-AI assistance group and Interpretable Joint-AI assistance group, their groups will be switched after a washout period.
Who Masked: Participant, Outcomes Assessor
Masking Description: During the endoscopic ultrasound procedure, the allocation of participants will be masked to the endoscopists
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Conventional diagnosis (No Intervention): Endoscopists diagnose pancreatic solid lesions according to endoscopic ultrasound images and clinical data.
- Joint-AI assisted diagnosis (Experimental): Endoscopists diagnose pancreatic solid lesions based on endoscopic ultrasound images, clinical data, and predictions made by the Joint-AI model.
  Interventions: Diagnostic Test: The assistance of the Joint-AI model
- Interpretable Joint-AI assisted diagnosis (Experimental): Endoscopists diagnose pancreatic solid lesions based on endoscopic ultrasound images, clinical data, predictions given by the Joint-AI, and interpretability analysis results used to improve the transparency of the decision-making process of the Joint-AI model.
  Interventions: Diagnostic Test: The assistance of the interpretable Joint-AI model

INTERVENTIONS:
Diagnostic Test: The assistance of the Joint-AI model — Predictions given by the Joint-AI model will be provided to the endoscopists during their diagnosis
  Arms: Joint-AI assisted diagnosis
Diagnostic Test: The assistance of the interpretable Joint-AI model — Predictions given by the Joint-AI model and the results of the interpretability analysis will be provided to the endoscopists during their diagnosis
  Arms: Interpretable Joint-AI assisted diagnosis

SUMMARY:
This clinical trial aims to learn if a multimodal artificial intelligence (AI) model can enhance the diagnosis of pancreatic solid lesions. The main questions it aims to answer are:

1. Does the AI model enhance the diagnostic performance of endoscopists in diagnosing pancreatic solid lesions?
2. Does the addition of interpretability analysis further improve the diagnostic performance of the assisted endoscopists? Researchers will compare the diagnostic performance of endoscopists with or without the assistance of the AI model.

Participants will:

1. Their clinical data will be prospectively collected.
2. They will be randomized to the AI-assist group and the conventional diagnosis group.

DETAILED DESCRIPTION:
The investigators have previously developed a multimodal AI model (Joint-AI) based on endoscopic ultrasound images and clinical data to diagnose pancreatic solid lesions. This study aims to improve the Joint-AI model's performance with a prospectively collected dataset and validate it through a randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Imaging examinations (MRI, CT, B-ultrasound) show a solid mass in the pancreas, which requires endoscopic ultrasound guided-fine needle aspiration/biopsy (EUS-FNA/B) to clarify the nature of the lesion in patients.
* Written consent provided

Exclusion Criteria:

* Age under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of correct diagnostic classification with assistance of the Joint-AI Model | Through study completion, an average of 1 year
  The rate of correct diagnoses in discriminating pancreatic cancer from other non-cancer lesions, determined by comparing endoscopist diagnosis assisted by the Joint-AI model against the final histopathological diagnosis (reference standard).
Rate of correct diagnostic classification with assistance of the Interpretable Joint-AI Model | Through study completion, an average of 1 year
  The rate of correct diagnoses in discriminating pancreatic cancer from other non-cancer lesions, determined by comparing endoscopist assessments assisted by the Interpretable Joint-AI model against the final histopathological diagnosis (reference standard)

SECONDARY OUTCOMES:
Rate of correct diagnostic classification of the Joint-AI model and the interpretable Joint-AI model | Through study completion, an average of 1 year
  Diagnostic accuracy of the AI models in this prospectively collected dataset.
Endoscopist-reported confidence score in diagnosis with AI assistance (the score is on a scale of 0%-100%, where 0 represents "not confident at all" and 100 represents "completely confident") | Through study completion, an average of 1 year
  Endoscopist-reported confidence in diagnosis will be measured on a scale ranging from 0 to 100, where 0 represents "not confident at all" and 100 represents "completely confident." Higher scores indicate greater diagnostic confidence. The confidence scores will be assessed separately for diagnoses made using the Joint-AI model and the interpretable Joint-AI model.
Rate of correct diagnostic classification of endoscopists without AI assistance | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China